CLINICAL TRIAL: NCT04078724
Title: Impact of Nutritional Supplementation on Gut-brain Axis in Older Adults With Normal Cognition vs. Mild Cognitive Impairment
Brief Title: Impact of Nutritional Supplementation on Sleep Quality and Gut Microbiome Composition in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Jung Eun Kim, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: S8
Record Dates: First submitted 2019-08-22; First posted 2019-09-06 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Sleep; Gut Microbiome
Keywords: Nutritional supplementation; Sleep quality; Cognitive function; Gut microbiome
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — 5-Hydroxytryptophan

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal subject without 5-HTP (Active Comparator): Subjects with normal cognition will be randomly assigned to not consuming 5-HTP.
  Interventions: Other: Without 5-HTP
- Normal subject with 5-HTP (Experimental): Subjects with normal cognition will be randomly assigned to consuming 100 mg of 5-HTP.
  Interventions: Dietary Supplement: 5-HTP

INTERVENTIONS:
Dietary Supplement: 5-HTP — 5-HTP that have Good Manufacturing Practice certification will be used and participants will be suggested to be take the 5-HTP supplementation at bedtime.
  Arms: Normal subject with 5-HTP
Other: Without 5-HTP — Subject will not take 5-HTP
  Arms: Normal subject without 5-HTP

SUMMARY:
The aim of this study is to assess the impact of 5-hydroxytryptophan (5-HTP) supplementation on sleep quality and gut microbiome composition in older adults with normal cognition vs. mild cognitive impairment (MCI) using a randomized controlled trial.

DETAILED DESCRIPTION:
This is a 12-wk parallel, single-bind (investigator), prospective study design with subjects randomly assigned to consume 100 mg of 5-HTP or does not consume 5-HTP. Fifty older men and women (aged 60-85y, approximately half men and half women, approximately half subjects with MCI) will be recruited with the expectation that ≥ 40 subjects (≥ 10 subjects per group) will complete the study. Body size, blood pressure, urinary melatonin, sleep quality, cognitive function and mood (including depression and anxiety), gut microbiome, and short chain fatty acids will be assessed. Blood amino acid concentration will be measured as an indicator of compliance to the 5-HTP consumption from the collected blood samples.

Relevance to Singapore: The results from the proposed research will assist a practical guidance of nutritional behavior changes providing gut and brain health promoting effects to Singapore older individuals with or without MCI and may result in reducing cost and manpower for cognitive decline care.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give an informed consent
2. Age 60 ≤years ≤ 85 years old
3. Weight change < 3kg in the past 3 months
4. Not exercising vigorously over the past 3 months
5. Not taking protein (e.g. Whey isolate, Ensure), tryptophan, serotonin and/or 5-HTP supplements for the past one month
6. Not taking sleep medication and/or dietary supplements for sleep (e.g. melatonin, GABA) for the past one month
7. Not taking prebiotic, probiotic and/or dietary fiber supplementations for the past one month
8. Not taking cognitive/brain supplementations (e.g. gingko biloba, acetylcholine) for the past one month
9. Not taking prescription anti-depressant or pain medication (e.g. Zoloft, Tramadol etc.)
10. No acute illness
11. If taking antihypertensive/cholesterol-lowering/ type 2 diabetic medication, he/she has been taking the medication for more than 5 years prior to the study participation
12. Not smoking
13. Not drinking more than 2 alcoholic drinks per day

Exclusion Criteria:

1. Unable to give an informed consent
2. Age < 60 years and >85 years old
3. Weight change >3kg in the past 3 months
4. Exercises vigorously over the past 3 months
5. Taking protein (e.g. Whey isolate, Ensure), tryptophan, serotonin and/or 5-HTP supplements for the past one month
6. Taking sleep medication and/or dietary supplements for sleep (e.g. melatonin, GABA) for the past one month
7. Taking prebiotic, probiotic and/or dietary fiber supplementations for the past one month
8. Taking cognitive/brain supplementation (e.g. gingko biloba, acetylcholine) for the past one month
9. Taking prescription anti-depressant or pain medication (e.g. Zoloft, Tramadol etc.)
10. Having acute illness
11. If taking antihypertensive/cholesterol-lowering/ type 2 diabetic medication, he/she has NOT been taking the medication for less than 5 years prior to the study participation
12. Smoking
13. Drinking more than 2 alcoholic drinks/day

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-07-04 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in sleep quality assessed by validated sleep questionnaires | Every 4 weeks (week 0, week 4, week 8 and week 12)
  Pittsburgh Sleep Quality Index Questionnaire (PSQI) will be used to assess the sleep quality. Overall score ranging from 0 to 21 points, where lower scores denote a healthier sleep quality.
Change in sleep quality assessed by electronic equipment | Every 4 weeks (week 0, week 4, week 8 and week 12)
  An electronic equipment, actigraphy, will be used to assess the sleep quality, including sleep timing and wake up timing.
Change in fecal short chain fatty acid (SCFA) concentration as assessed by micromoles per gram (μmol/g) | Pre- and post-intervention (week 0 and week 12)
  Fecal SCFA concentration will be measured using gas chromatograph (GC) and assessed by μmol/g. There is no recognized range. Normally the higher level is better.
Change in fecal microbiome composition | Pre- and post-intervention (week 0 and week 12)
  High-throughput sequencing method (using Illumina MiSeq platforms) will be used to assess the changes in gut microbiome composition.

SECONDARY OUTCOMES:
Change in Quality of Life: WHOQOL | Every 4 weeks (week 0, week 4, week 8 and week 12)
  The World Health Organization Quality of Life Assessment (WHOQOL) will be used to assess the quality of life. Score ranging from 0 to 100 points, where higher scores denote higher quality of life.
Change in Cognitive function | Every 4 weeks (week 0, week 4, week 8 and week 12)
  Montreal Cognitive Assessment (MOCA) will be used to assess the cognitive function. Score ranging from 0 to 30 points. A final total score of 26 and above is considered normal.
Change in mood (depression) | Every 4 weeks (week 0, week 4, week 8 and week 12)
  Geriatric Depression Scale (GDS) Assessment will be used to assess the depression situation. Score ranging from 0 to 15 points. Although differing sensitivities and specificities have been obtained across studies, for clinical purposes a score > 5 points is suggestive of depression and should warrant a follow-up interview. Scores > 10 are almost always depression.
Change in mood (anxiety) | Every 4 weeks (week 0, week 4, week 8 and week 12)
  Geriatric Anxiety Inventory (GAI) Assessment will be used to assess the anxiety situation. Score ranging from 0 to 20 points, where higher scores denote higher level of anxiety.
Change in urinary melatonin levels as assessed by nanogram per milliliter (ng/mL) | Pre- and post-intervention (week 0 and week 12)
  Change in urinary melatonin levels will be assessed by using enzyme linked immunosorbent assay (ELISA) kits. There is no recognized range. Normally the higher level is better.
Change in blood amino acids assessed by nanomole per milliliter (ng/mL) | Pre- and post-intervention (week 0 and week 12)
  Amino Acid Analysis System will be used to assess the blood amino acid levels. There is no recognized range.
Change in weight and height | Every 4 weeks (week 0, week 4, week 8 and week 12)
  Weight (in kilograms) and height (in meters) will be combined to report BMI in kg/m^2.
Change in waist circumference as assessed by centimeter (cm) | Every 4 weeks (week 0, week 4, week 8 and week 12)
  Recommended cutoffs for increased health risk are a waist circumference >102 cm for men and >88 cm for women.
Dietary assessment | Every 4 weeks (week 0, week 4, week 8 and week 12)
  Dietary assessment will be assessed by 3-day dietary food record.
Blood pressure as assessed by millimeter of mercury (mmHg) | Every 4 weeks (week 0, week 4, week 8 and week 12)
  Systolic and diastolic blood pressure will be measured by a blood pressure monitor. For a normal reading, systolic pressure is between 90 and 120 and diastolic pressure is between 60 and 80.

CONTACTS AND LOCATIONS:
Overall Officials: Kim J Eun, PhD, Principal Investigator — National University of Singapore
Locations (2):
- Singapore (2):
  - National University of Singapore, Singapore
  - Hannah Seniors Activity Centre, Singapore

IPD SHARING:
Plan to Share IPD: No
Electronic copies of the data with identifiable participant information will be kept on a secure website with access limited to Dr. Kim and her research staff. All data will be de-identified prior to statistical analyses

REFERENCES:
- [Background] Mohajeri MH, Wittwer J, Vargas K, Hogan E, Holmes A, Rogers PJ, Goralczyk R, Gibson EL. Chronic treatment with a tryptophan-rich protein hydrolysate improves emotional processing, mental energy levels and reaction time in middle-aged women. Br J Nutr. 2015 Jan 28;113(2):350-65. doi: 10.1017/S0007114514003754. Epub 2015 Jan 9. PMID 25572038
- [Result] Anderson JR, Carroll I, Azcarate-Peril MA, Rochette AD, Heinberg LJ, Peat C, Steffen K, Manderino LM, Mitchell J, Gunstad J. A preliminary examination of gut microbiota, sleep, and cognitive flexibility in healthy older adults. Sleep Med. 2017 Oct;38:104-107. doi: 10.1016/j.sleep.2017.07.018. Epub 2017 Aug 2. PMID 29031742
- [Derived] Sutanto CN, Xia X, Heng CW, Tan YS, Lee DPS, Fam J, Kim JE. The impact of 5-hydroxytryptophan supplementation on sleep quality and gut microbiota composition in older adults: A randomized controlled trial. Clin Nutr. 2024 Mar;43(3):593-602. doi: 10.1016/j.clnu.2024.01.010. Epub 2024 Jan 17. PMID 38309227